CLINICAL TRIAL: NCT00242099
Title: The Clinical Utility of Monitoring for Human Herpesvirus-6 (HHV-6) and Human Herpesvirus-7 (HHV-7) After Liver Transplant: A Randomized Trial
Brief Title: Clinical Utility of Monitoring for Human Herpesvirus-6 (HHV-6) and Human Herpesvirus-7 (HHV-7) After Liver Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 04-0760-AE; PSI-04-53
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2005-02

CONDITIONS: Transplant
Keywords: liver transplant; HHV-6; HHV-7; Human Herpesvirus-6; Human Herpesvirus-7

INTERVENTIONS:
Procedure: Monitoring - blood samples drawn to test for HHV-6 and HHV-7

SUMMARY:
Human herpesvirus-6 (HHV-6) and -7 (HHV-7) infections are common after transplantation. Such infections may predispose transplant patients to other infections, contribute to a recurrence of hepatitis C virus, and affect rejection and function of the transplanted liver. Given the significant clinical impact of these viruses, routine laboratory monitoring may be beneficial by identifying patients who have persistent or high levels of infection. In these patients, immunosuppressive medications could be adjusted, or antiviral medications administered. There are currently no randomized trials that address this important question. This prospective, randomized trial will analyze whether routine laboratory monitoring for HHV-6 and -7 is clinically useful, and whether it would improve overall outcomes in transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who fulfill the following criteria are eligible for inclusion:

  * Recipients of a liver transplant
  * Able to give written informed consent
  * Are willing and able to comply with the protocol
  * Age >= 18 years

Exclusion Criteria:

The following patients are not eligible for inclusion in the study:

* Patients unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Adverse clinic events due to direct or indirect effects.

CONTACTS AND LOCATIONS:
Overall Officials: Atul Humar, MD, Principal Investigator — University Health Network, Toronto; Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Fernandez-Ruiz M, Kumar D, Husain S, Lilly L, Renner E, Mazzulli T, Moussa G, Humar A. Utility of a monitoring strategy for human herpesviruses 6 and 7 viremia after liver transplantation: a randomized clinical trial. Transplantation. 2015 Jan;99(1):106-13. doi: 10.1097/TP.0000000000000306. PMID 25073037